CLINICAL TRIAL: NCT02975700
Title: A Phase I/II Open Label, Multicenter Study of PLX3397 in Patients With Unresectable or Metastatic KIT-mutated Melanoma
Brief Title: A Study of PLX3397 in Patients With Unresectable or Metastatic KIT-mutated Melanoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-13
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: PLX3397; Kit-mutant Melanoma; Unresectable or Metastatic KIT-mutated Melanoma; Developmental Phase I/II
MeSH Terms: conditions — Melanoma | interventions — pexidartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PLX3397 (Experimental): Part 1: Open label, multicenter study includes a dose evaluation portion in which the safety profile of PLX3397 as a single oral agent will be evaluated
  Part 2: An expansion cohort in which the efficacy and safety of PLX3397 administered at the recommended Phase 2 dose will be evaluated in patients with unresectable stage III or stage IV KIT-mutated melanoma.
  Interventions: Drug: PLX3397

INTERVENTIONS:
Drug: PLX3397 — 1000 mg/day (400 mg in the morning and 600 mg in the evening)
  Other Names: Pexidartinib

SUMMARY:
The purpose of this Phase I/II study is to evaluate safety, pharmacokinetics, and preliminary efficacy of the investigational drug PLX3397 in subjects with unresectable or metastatic KIT-mutated melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unresectable stage III or stage IV melanoma which is histologically confirmed at the treating institution with KIT mutation(s) not known to be resistant to PLX3397
* Presence of measurable lesions by Response Evaluation Criteria in Solid Tumors
* Eastern Cooperative Oncology Group (ECOG) performance Status (PS) 0-2
* Life expectancy ≥ 3 months
* Adequate organ and bone marrow function
* Women of child-bearing potential must have a negative serum pregnancy test at Screening and must agree to use an effective form of contraception from the time of the negative pregnancy test up to 3 months after the last dose of study drug. Women of non-child-bearing potential must have been postmenopausal for ≥ 1 year or surgically sterile.
* Fertile men must agree to use an effective method of birth control during the study and for up to 3 months after the last dose of study drug.
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements

Exclusion Criteria:

* Prior treatment with a KIT inhibitor for melanoma
* Presence of NRAS or BRAF mutation
* Exposure to any investigational drug within 28 days or unresolved adverse effects from previous therapy
* Symptomatic brain metastases.
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Sponsor
* Concomitant treatment with other anti-neoplastic agents (hormonal therapy acceptable)
* Uncontrolled intercurrent or infectious illness
* Major surgical procedure or significant traumatic injury within 14 days of initiating study drug or anticipation of the need for major surgery during the study
* Previous radiotherapy to 25% or more of the bone marrow and/or radiation therapy within 28 days prior to study entry
* Inability to swallow capsules, or refractory nausea and vomiting, malabsorption, an external biliary shunt, or significant bowel resection that would preclude adequate absorption
* Congestive heart failure (CHF) New York (NY) Heart Association class III or IV; unstable coronary artery disease [myocardial infarction (MI) more than 6 months prior to study entry is permitted] or serious cardiac arrhythmia
* Baseline QT interval corrected using Fridericia equation (QTcF) ≥ 450 msec (for males) or ≥ 470 msec (for females) at Screening
* Active or chronic infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV)
* Known chronic liver disease
* Women who are breast-feeding or pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2024-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (5):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen Hospital, Guangzhou, Guangdong
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-Gu
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants entered the pilot portion of the study; no participants entered the phase 2 portion. Of the 8 participants, 2 failed screening criteria and did not receive treatment.
Groups:
- PLX3397: Participants who received PLX3397 1000 mg/day (400 mg in the morning and 600 mg in the evening).
Period: Overall Study
Arm/Group | PLX3397
Started | 6
Completed | 0
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Progressive disease | 3
Not completed — Failed screening criteria | 2

BASELINE CHARACTERISTICS:
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 6

OUTCOME MEASURES:

1. Primary Outcome: Summary of Best Overall Response Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: For the assessment of best overall response, participants were classified by RECIST v1.1: complete response (CR), disappearance of all target lesions and normalization of tumor marker level; partial response (PR), at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters; stable disease (SD); neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study; progressive disease (PD), at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm; or not evaluable (NE) for analysis.
Time Frame: within 18 months postdose
Population: Best overall response was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Complete response (CR) | 0
  Partial response (PR) | 1
  Stable disease (SD) | 2
  Progressive disease (PD) | 1
  Not evaluable (NE) | 2

2. Primary Outcome: Objective Response Rate (ORR) Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Objective response rate was defined as complete response (CR) or partial response (PR).
Time Frame: within 18 months postdose
Population: Objective response rate among participants who achieved complete response or partial response was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants | 1

3. Secondary Outcome: Duration of Response Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Duration of Response (DoR) was defined as the time from the first documentation of objective tumor response (complete response [CR] or partial response [PR]) to the first documentation of disease progression or to death due to any cause, whichever occurred first. DoR was to only be calculated for the subgroup of participants with an objective tumor response.
Time Frame: within 18 months postdose
Population: Duration of response was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Median (Full Range); unit: months
Arm/Group | PLX3397
Number analyzed (Participants) | 1
months | NA [8.15 to 8.15] — Lack of a median value is due to fewer than 50% of the participants experiencing the event.

4. Secondary Outcome: Progression-free Survival Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Progression-free survival (PFS) was to be calculated for each participant as the number of days from study enrollment to the date of the first documented disease progression or date of death from any cause, whichever occurred first.
Time Frame: within 18 months postdose
Population: Progression-free survival was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PLX3397
Number analyzed (Participants) | 6
months | 10.32 [1.58 to NA] — Missing upper bound is related to right-censored data. Last time point censored and estimate is essentially infinity, therefore it is NA.

5. Secondary Outcome: Overall Survival Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Overall survival (OS) was defined as the time from study enrollment to death from any cause, censoring at the date of last contact or the end of the study.
Time Frame: within 18 months postdose
Population: Overall survival was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | PLX3397
Number analyzed (Participants) | 6
months | NA [4.11 to NA] — There were not enough events to estimate the median survival time.

6. Secondary Outcome: Disease Control Rate Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Disease control rate (DCR) was defined as the percentage of participants who had achieved complete response (CR), partial response (PR), or stable disease (SD).
Time Frame: within 18 months postdose
Population: Disease control rate among participants who achieved CR, PR, or SD was assessed in the Modified Intent-to-Treat Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants | 3

7. Secondary Outcome: Summary of Pharmacokinetic Parameter of Maximum Concentration (Cmax) of PL3397 at Days 1 and 15 Following Twice Daily Administration of PL3397 at 1000 mg/Day in Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5 h, 1h, 2h, 4h, and 6h postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PLX3397
Number analyzed (Participants) | 6
ng/mL
  Day 1 | 4660 (1830)
  Day 15: number analyzed (Participants) | 5
  Day 15 | 9570 (2940)

8. Secondary Outcome: Summary of Pharmacokinetic Parameter of Area Under the Curve From Zero to 6 Hours (AUC0-6) of PL3397 at Days 1 and 15 Following Twice Daily Administration of PL3397 at 1000 mg/Day in Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5 h, 1h, 2h, 4h, and 6h postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | PLX3397
Number analyzed (Participants) | 6
h*ng/mL
  Day 1 | 14500 (4660)
  Day 15: number analyzed (Participants) | 5
  Day 15 | 43800 (7010)

9. Secondary Outcome: Summary of Pharmacokinetic Parameter of Time to Maximum Concentration and Last Measurable Time of PL3397 at Days 1 and 15 Following Twice Daily Administration of PL3397 at 1000 mg/Day in Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5 h, 1h, 2h, 4h, and 6h postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PLX3397
Number analyzed (Participants) | 6
hours
  Time to maximum concentration; Day 1 | 2.72 (1.62)
  Time to maximum concentration; Day 15: number analyzed (Participants) | 5
  Time to maximum concentration; Day 15 | 2.77 (2.31)
  Last measurable time; Day 1 | 5.99 (0.05)
  Last measurable time; Day 15: number analyzed (Participants) | 5
  Last measurable time; Day 15 | 6.03 (0.06)

10. Secondary Outcome: Summary of Pharmacokinetic Parameter of Accumulation Ratio of Day 15 to Day 1 for AUC0-6h (Robs) of PL3397 at Day 15 Following Twice Daily Administration of PL3397 at 1000 mg/Day in Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5 h, 1h, 2h, 4h, and 6h postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PLX3397
Number analyzed (Participants) | 5
Ratio | 3.39 (0.85)

11. Secondary Outcome: Summary of Pharmacokinetic Parameter of Accumulation Ratio of Day 15 to Day 1 for Cmax (Rcmax) of PL3397 at Day 15 Following Twice Daily Administration of PL3397 at 1000 mg/Day in Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: Cycle 1, Day 1 and Day 15 at predose, 0.5 h, 1h, 2h, 4h, and 6h postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | PLX3397
Number analyzed (Participants) | 5
Ratio | 2.34 (0.69)

12. Secondary Outcome: Summary of Most Common (≥50% of Participants) Treatment-emergent Adverse Events Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: within 28 days after administration of the last dose of study drug, up to 18 months postdose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Aspartate aminotransferase increased | 6
  White blood cell count decreased | 6
  Anaemia | 5
  Face oedema | 5
  Alanine aminotransferase increased | 4
  Blood bilirubin increased | 4
  Gamma-glutamyltransferase increased | 4
  Hair colour changes | 4
  Neutrophil count decreased | 4
  Bilirubin conjugated increased | 3
  Blood alkaline phosphatase increased | 3
  Blood lactate dehydrogenase increased | 3
  Interstitial lung disease | 3
  Pyrexia | 3
  Total bile acids increased | 3

13. Secondary Outcome: Summary of Treatment-emergent Adverse Events Grade ≥ 3 Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: Grade ≥ 3 was used to indicate moderate-to-severe treatment-emergent adverse events in which moderate was defined as discomfort enough to cause interference with normal daily activities and severe defined as the inability to perform normal daily activities.
Time Frame: within 28 days after administration of the last dose of study drug, up to 18 months postdose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Any TEAEs CTCAE Grade ≥ 3 | 4
  Gamma-glutamyltransferase increased | 4
  Alanine aminotransferase increased | 2
  Total bile acids increased | 2
  Anaemia | 1
  Aspartate aminotransferase increased | 1
  Bilirubin conjugated increased | 1
  Blood alkaline phosphatase increased | 1
  Blood bilirubin increased | 1
  Drug-induced liver injury | 1
  Herpes zoster | 1
  Hypertension | 1
  Neutrophil count decreased | 1
  White blood cell count decreased | 1

14. Secondary Outcome: Summary of Most Common (≥50%) Drug-related Treatment-emergent Adverse Events Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Time Frame: within 28 days after administration of the last dose of study drug, up to 18 months postdose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Aspartate aminotransferase increased | 6
  White blood cell count decreased | 6
  Anaemia | 5
  Face oedema | 5
  Alanine aminotransferase increased | 4
  Blood bilirubin increased | 4
  Gamma-glutamyltransferase increased | 4
  Hair colour changes | 4
  Neutrophil count decreased | 4
  Bilirubin conjugated increased | 3
  Blood alkaline phosphatase increased | 3
  Blood lactate dehydrogenase increased | 3
  Interstitial lung disease | 3
  Total bile acids increased | 3

15. Secondary Outcome: Summary of Drug-related Treatment-emergent Adverse Events Grade ≥ 3 Following Twice Daily Administration of PL3397 at 1000 mg/Day In Participants With Unresectable or Advanced KIT-mutated Melanoma
Description: as for outcome 13
Time Frame: within 28 days after administration of the last dose of study drug, up to 18 months postdose
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | PLX3397
Number analyzed (Participants) | 6
Participants
  Any Drug-related TEAEs CTCAE Grade ≥ 3 | 4
  Gamma-glutamyltransferase increased | 4
  Alanine aminotransferase increased | 2
  Total bile acids increased | 2
  Aspartate aminotransferase increased | 1
  Bilirubin conjugated increased | 1
  Blood alkaline phosphatase increased | 1
  Blood bilirubin increased | 1
  Drug-induced liver injury | 1
  Neutrophil count decreased | 1
  White blood cell count decreased | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from after initiation of study drug up to 28 days after administration of last dose of study drug, up to 18 months postdose.
Arm/Group | PLX3397
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=6)
Drug-induced liver injury (Hepatobiliary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PLX3397 (N=6)
Face oedema (General disorders) | 5
Pyrexia (General disorders) | 3
Fatigue (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 6
White blood cell count decreased (Investigations) | 6
Alanine aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 3
Gamma-glutamyltransferase increased (Investigations) | 4
Neutrophil count decreased (Investigations) | 4
Bilirubin conjugated increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 3
Total bile acids increased (Investigations) | 3
Red blood cell count decreased (Investigations) | 4
Blood creatinine phosphokinase increased (Investigations) | 2
Blood potassium decreased (Investigations) | 1
Blood triglycerides increased (Investigations) | 1
Blood urea increased (Investigations) | 2
Blood uric acid increased (Investigations) | 1
Creatinine renal clearance decreased (Investigations) | 2
Electrocardiogram QT prolonged (Investigations) | 1
Glucose urine present (Investigations) | 2
Urine ketone body present (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 6
Hair colour changes (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Eyelid oedema (Eye disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Hypertension (Vascular disorders) | 1
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 2
Blood chloride decreased (Investigations) | 2
Blood cholesterol increased (Investigations) | 2
Blood creatine phosphokinase MB increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
High density lipoprotein increased (Investigations) | 2
Low density lipoprotein increased (Investigations) | 2
Albumin globulin ratio increased (Investigations) | 1
Blood magnesium increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Electrocardiogram high voltage (Investigations) | 1
Electrocardiogram ST-T change (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Mean cell volume abnormal (Investigations) | 1
Protein urine present (Investigations) | 1
Urobilinogen urine increased (Investigations) | 1
White blood cells urine positive (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Corona virus infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Amnesia (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Cervical polyp (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT02975700/Prot_SAP_000.pdf